CLINICAL TRIAL: NCT00013962
Title: Vitamin D Metabolism and the Williams Syndrome
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Other Study IDs: NCRR-M01RR01070-0562
Record Dates: First submitted 2001-04-03; First posted 2001-04-05 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Williams Syndrome
MeSH Terms: conditions — Williams Syndrome | interventions — Vitamin D

STUDY DESIGN:
Observational Model: Case-Control

INTERVENTIONS:
Drug: Vitamin D

SUMMARY:
The Williams syndrome is a disease in which supravalvular aortic stenosis, an elfin facies, mental retardation and other congenital defects are sometimes associated with abnormal vitamin D and calcium metabolism. Whereas some patients have been reported to show increased sensitivity to vitamin D or an exaggerated response of serum 25-hydroxyvitamin D {25(OH)D} to administration of vitamin D and to have hypercalcemia caused by increased circulating 1,25-dihydroxyvitamin D{1,25(OH)2D} in infancy and early childhood, most patients have normal calcium metabolism and normal values for circulating 25(OH)D and 1,25(OH)2D. We propose to carry out further studies of vitamin D metabolism to elucidate the mechanism(s) for abnormal vitamin D metabolism. We will determine the response of serum 1,25(OH)2D to administration of 1,25(OH)2D3. Measurement of the 1,25(OH)2D in the patients compared to normal subjects will be the primary outcome.

ELIGIBILITY:
Age 18 years to 50 years of age, patients and normal subjects

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States